CLINICAL TRIAL: NCT03020953
Title: The Anabolic Effects of Estrogen on Skeletal Muscles
Acronym: ESTRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Estrogen2016
Record Dates: First submitted 2016-12-15; First posted 2017-01-13 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2018-06

CONDITIONS: Estrogen Supplementation
MeSH Terms: interventions — Exercise; Estrogens

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise + Estrogen (Experimental): Strength training 3 times a week for 12 weeks. Estrogen patches which provide 100 um pr. 24 hours.
  Interventions: Other: Exercise + Estrogen
- Exercise + Placebo (Active Comparator): Strength training 3 times a week for 12 weeks. Placebo patches.
  Interventions: Other: Exercise + Placebo

INTERVENTIONS:
Other: Exercise + Estrogen — 12 weeks resistance training and estrogen patches
  Arms: Exercise + Estrogen
Other: Exercise + Placebo — 12 weeks resistance training and placebo patches
  Arms: Exercise + Placebo

SUMMARY:
Purpose: to study the effect of estrogen replacement on muscle hypertrophy in response to 12 weeks resistance training in postmenopausal women Hypothesis: Transdermal administration of 17-β estradiol enhance the anabolic effect of resistance training on muscle mass, strength in postmenopausal women Primary outcome: Muscle hypertrophy (muscle CSA, muscle fiber type specific CSA) Secondary outcome: Messenger RiboNucleic Acid (mRNA)(real-time PCR), protein (western blotting), satellite cell proliferation and activation, Strength, functional test, muscle protein synthese.

Design: Two groups of healthy postmenopausal women (½-5 years after menopause) who have not performed regular resistance exercise (<1 times per week) the last two years. Randomized, controlled intervention study +/- transdermal administration of estrogen (17-β estradiol). Both groups perform 12 weeks of supervised progressive resistance training (3/week) aiming to induce muscle hypertrophy in the legs.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, more than 6 months, but less than 5 years since last menstruation.

Exclusion Criteria:

* Less than 2 hours exercise with moderate to high intensity per week the last year, no regular resistance exercise the last 2 years (less than 5 exercise bouts during the last year)
* No previous or present lower limb injuries which may hinder participation in strength training
* No use of medicine which may influence the adaptation to strength training such as regular use of nonsteroidal anti-inflammatory drugs and use of statins, no muscle
* Joint or metabolic diseases or other chronic diseases that would affect the results of the investigation, high blood pressure (>140/90), smoking

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Muscle hypertrophy | 12 weeks
  muscle cross sectional area measured by Magnetic resonance imaging (MR) -scans

SECONDARY OUTCOMES:
Muscle fiber hypertrophy | 12 weeks
  Histology analysis of muscle fiber area
Muscle strength | 12 weeks
  Maximal isometric muscle strength
tendon size | 12 weeks
  Tendon cross sectional area measured by MR-scan
Fat cell size | 12 weeks
  Analysis of fat cell size (diameter)
Fat mass | 12 weeks
  Dual-energy X-ray absorptiometry (DXA) scan of total fat mass
Fat free mass | 12 weeks
  Fat free mass measured by DXA scan

CONTACTS AND LOCATIONS:
Overall Officials: Mette Hansen, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Sport Science, Department of Public Health, Aarhus University, Aarhus, Denmark

REFERENCES:
- [Derived] Dam TV, Dalgaard LB, Johansen FT, Bengtsen MB, Mose M, Lauritsen KM, Gravholt CH, Hansen M. Effects of transdermal estrogen therapy on satellite cell number and molecular markers for muscle hypertrophy in response to resistance training in early postmenopausal women. Eur J Appl Physiol. 2023 Mar;123(3):667-681. doi: 10.1007/s00421-022-05093-0. Epub 2022 Dec 31. PMID 36585491